CLINICAL TRIAL: NCT02595944
Title: Adjuvant Nivolumab in Resected Lung Cancers (ANVIL)-A Randomized Phase III Study of Nivolumab After Surgical Resection and Adjuvant Chemotherapy in Non-Small Cell Lung Cancers
Brief Title: Nivolumab After Surgery and Chemotherapy in Treating Patients With Stage IB-IIIA Non-small Cell Lung Cancer (An ALCHEMIST Treatment Trial)
Acronym: ANVIL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01916; NCI-2015-01916 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); s16-02074; EA5142 (Other: ECOG-ACRIN Cancer Research Group); EA5142 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Stage IB Lung Non-Small Cell Carcinoma AJCC v7; Stage II Lung Non-Small Cell Cancer AJCC v7; Stage IIIA Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Specimen Handling; Nivolumab; Observation; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 4 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or PET/CT throughout the trial and blood sample collection during screening and follow-up. Patients may undergo an ECHO as clinically indicated on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Biological: Nivolumab; Procedure: Positron Emission Tomography
- Arm II (observation) (Active Comparator): Patients are followed serially with CT and/or PET/CT imaging for up to 1 year and then during follow-up. Patients also undergo blood sample collection during screening and follow-up. Patients may undergo an ECHO as clinically indicated on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Other: Observation Activity; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm I (nivolumab)
Other: Observation Activity — Undergo observation
  Other Names: Observation
  Arms: Arm II (observation)
Procedure: Positron Emission Tomography — Undergo PET-CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase III ALCHEMIST treatment trial studies how well nivolumab after surgery and chemotherapy work in treating patients with stage IB-IIIA non-small cell lung cancer. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether adjuvant therapy with nivolumab will result in improved disease-free survival (DFS) over standard observation in patients with stage IB >= 4 cm, II and IIIA, non-small cell lung cancer (NSCLC) following surgical resection and standard adjuvant therapy.

II. To evaluate whether adjuvant therapy with nivolumab will result in improved disease-free survival (DFS) over standard observation in patients with stage IB >= 4cm, II and IIIA, NSCLC with high PD-L1 expression (>= 50% staining) following surgical resection and standard adjuvant therapy.

III. To evaluate whether adjuvant therapy with nivolumab will result in improved overall survival (OS) over standard observation in patients with stage IB >= 4cm, II and IIIA, NSCLC following surgical resection and standard adjuvant therapy.

SECONDARY OBJECTIVES:

I. To evaluate the safety profile of nivolumab when given as an adjuvant therapy.

II. To evaluate and compare disease free and overall survival in patients with tumors that express PD-L1 in various patterns associated with nivolumab and standard observation.

III. To evaluate and compare disease free and overall survival in patients with tumors that have high mutational load associated with nivolumab and standard observation.

IV. To evaluate OS and DFS by stage. V. To evaluate OS and DFS by each stratification factor.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 4 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and/or positron emission tomography (PET)/CT throughout the trial and blood sample collection during screening and follow-up. Patients may undergo an echocardiography (ECHO) as clinically indicated on study.

ARM II: Patients are followed serially with CT and/or PET/CT imaging for up to 1 year and then during follow-up. Patients also undergo blood sample collection during screening and follow-up. Patients may undergo an ECHO as clinically indicated on study.

After completion of study treatment, patients are followed up at 6 weeks, every 3 months for 2 years, every 6 months for 2 years, and then every 12 months for 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Patients must have undergone complete surgical resection of their stage IB (>= 4 cm), II or IIIA NSCLC according to the American Joint Committee on Cancer (AJCC) 7th edition and have had negative surgical margins
* Baseline chest CT must be performed within 1 month (30 days) prior to randomization to ensure no evidence of disease; if clinically indicated, additional imaging studies must be performed to rule out metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients must be registered to the ALCHEMIST-SCREEN (ALLIANCE A151216) trial prior to randomization
* Non-squamous tumors must not be positive for EGFR exon 19 deletion or exon 21 L858R mutation (centrally as part of the ALCHEMIST-SCREEN protocol) and ALK rearrangement (centrally as part of ALCHEMIST-SCREEN and/or locally)

  * NOTE: if the results of the central EGFR testing are negative, but the ALK testing was not able to be completed by the ALCHEMIST central lab, the ALK status will be considered negative (unless locally positive for ALK rearrangement) and the patient may be considered for enrollment onto EA5142, once PD-L1 results are received and all other eligibility requirements are met
* Tumors must have PD-L1 status tested centrally as part of the ALCHEMIST-SCREEN protocol
* Women must not be pregnant or breast-feeding due to unknown and potentially harmful effects of nivolumab on the developing fetus or child
* All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception or to abstain from sexual intercourse during the treatment period and for 31 weeks after the last nivolumab infusion
* Patients must NOT have uncontrolled intercurrent illness including, but not limited to, serious ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements
* No prior treatment with an immune checkpoint inhibitor (anti-PD-1, anti-PD-L1, anti-CTLA4 monoclonal antibody)
* Patients must have adequately recovered from thoracic surgery and any administered chemotherapy/radiotherapy at the time of randomization (NOTE: adjuvant chemotherapy and/or radiation is not required)

  * Minimum time between date of surgery and randomization is 4 weeks (28 days)
  * Maximum time allowed between surgery and randomization:

    * 3 months (90 days) if no chemotherapy is administered
    * 8 months (240 days) if adjuvant chemotherapy was administered
    * 10 months (300 days) if adjuvant chemotherapy and radiation therapy was administered
* Patients must have completed and recovered from any adjuvant chemotherapy 2 or more weeks prior to randomization (6 weeks for mitomycin and nitrosoureas; 4 weeks for post-operative radiation therapy) (NOTE: adjuvant chemotherapy and/or radiation is not required)
* Serum aspartate transaminase (aspartate aminotransferase [AST]) and serum alanine transaminase (alanine aminotransferase [ALT]) =< 2.5 x upper limit normal (within 2 weeks prior to randomization)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (except in subjects with Gilbert syndrome who must have a total bilirubin < 3.0 x ULN) (within 2 weeks prior to randomization)
* White blood cell (WBC) >= 2000/uL (within 2 weeks prior to randomization)
* Neutrophils >= 1000/uL (within 2 weeks prior to randomization)
* Platelets >= 100 x 10^3/uL (within 2 weeks prior to randomization)
* Hemoglobin >= 8 g/dL (within 2 weeks prior to randomization)
* Serum creatinine =< 2 x ULN (within 2 weeks prior to randomization)
* Prior to randomization patients with any non-hematologic toxicity from surgery, chemotherapy and radiation therapy must have recovered to grade =< 1 with the exception of alopecia, ototoxicity and neuropathy
* Patients must not be receiving any other investigational anti-cancer agents while on study
* Patients must not have known or suspected autoimmune disease; subjects with type I diabetes mellitus, hypothyroidism requiring hormone replacement, or skin disorders not requiring systemic treatment are permitted to enroll
* Patients must not have a condition requiring systemic corticosteroids equivalent to > 10 mg prednisone per day or other immunosuppressive medications within 2 weeks of randomization; inhaled, intra-articular, and epidural steroids are permissible
* Patients must not have known interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Patients must not have a known history of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection that is untreated and/or with a detectable viral load
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 903 (Estimated)
Dates: Start 2016-07-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Time from randomization to the earliest event defined as disease recurrence, any new lung cancer (even in the opposite lung), or death from any cause at any known point in time, assessed up to 10 years
  DFS distributions will be estimated using the Kaplan-Meier method, and Cox proportional hazards models will be used to estimate the treatment hazard ratios. The primary comparisons of DFS will use a logrank tests stratified on the randomization stratification factors with a one-sided type I error rate corresponding to the significance level associated with population being analyzed; that is, 1.5% for the overall population and 1% for the >= 50% population. The latter test will only be performed in the event that the primary test in all-comers is not statistically significant. Other comparisons of groups will be made using the logrank test and Cox modeling. Point estimates of all endpoints will be accompanied by the corresponding confidence intervals adjusted for the type I error rates associated with the endpoint. Subset analyses are planned for all stratification factors and all known prognostic factors such as performance status, age, gender, etc.
Overall survival (OS) | From randomization to death from any cause, assessed up to 10 years
  OS distributions will be estimated using the Kaplan-Meier method, and Cox proportional hazards models will be used to estimate the treatment hazard ratios. The primary comparisons of OS will use a logrank tests stratified on the randomization stratification factors with a one-sided type I error rate corresponding to the significance level associated with population being analyzed; that is, 1.5% for the overall population and 1% for the >= 50% population. The latter test will only be performed in the event that the primary test in all-comers is not statistically significant. Other comparisons of groups will be made using the logrank test and Cox modeling. Point estimates of all endpoints will be accompanied by the corresponding confidence intervals adjusted for the type I error rates associated with the endpoint. Subset analyses are planned for all stratification factors and all known prognostic factors such as performance status, age, gender, etc.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 10 years
  Toxicity graded according to Common Terminology Criteria for Adverse Events version 5.0. Toxicity rates will be compared using Fisher's exact tests with a one-sided type I error rate of 2.5%; multivariable logistic regression modeling will be used to adjust for the effect of any covariates that are associated with these categorical outcomes. Point estimates of all endpoints will be accompanied by the corresponding confidence intervals adjusted for the type I error rates associated with the endpoint. Subset analyses are planned for all stratification factors and all known prognostic factors such as performance status, age, gender, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie E Chaft, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (886):
- United States (886):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Southern Cancer Center PC-Daphne, Daphne, Alabama
  - Southern Cancer Center PC-Mobile, Mobile, Alabama
  - Southern Cancer Center PC-Providence, Mobile, Alabama
  - Southern Cancer Center PC-Springhill, Mobile, Alabama
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Eden Hospital Medical Center, Castro Valley, California
  - University Oncology Associates, Clovis, California
  - John Muir Medical Center-Concord, Concord, California
  - City of Hope Corona, Corona, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Saint Jude Medical Center, Fullerton, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Mercy Regional Cancer Center, Redding, California
  - Mercy Oncology Center, Redding, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Dominican Santa Cruz Hospital, Santa Cruz, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Saint Helena Hospital, St. Helena, California
  - Saint Joseph's Medical Center, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - The Watson Clinic, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Indian River Medical Center, Vero Beach, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Quincy Medical Group-Clinic, Quincy, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - MercyOne Genesis Silvis Cancer Center, Silvis, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - The Community Hospital, Munster, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - MercyOne Genesis Davenport Medical Center, Davenport, Iowa
  - MercyOne Genesis Davenport Cancer Center, Davenport, Iowa
  - Iowa Cancer Specialists, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Iowa City VA Healthcare System, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - King's Daughter's Medical Center, Ashland, Kentucky
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - Saint Elizabeth Healthcare Fort Thomas, Fort Thomas, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - CHRISTUS Saint Patrick Hospital, Lake Charles, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - CHRISTUS Highland Medical Center, Shreveport, Louisiana
  - Ochsner Hematology Oncology North Shore - Slidell (East Region), Slidell, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - New England Cancer Specialists - Kennebunk, Kennebunk, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - New England Cancer Specialists - Topsham, Topsham, Maine
  - New England Cancer Specialists, Westbrook, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Boston Medical Center - Brighton, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - UP Health System Hematology Oncology Marquette, Marquette, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Forrest General Hospital / Cancer Center, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Veteran's Affairs Medical Center - Saint Louis, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - The Dana-Farber Cancer Institute at Londonderry, Londonderry, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newton Medical Center, Newton, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Chilton Medical Center, Pompton, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - Lovelace Medical Center-Downtown, Albuquerque, New Mexico
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Gaston Hematology and Oncology Associates, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Maria Parham Hospital, Henderson, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Scotland Memorial Hospital-Laurinburg Cancer Center, Laurinburg, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Johnston Memorial Hospital, Smithfield, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Toledo, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Good Samaritan Hospital, Corvallis, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Family Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Hendrick Medical Center, Abilene, Texas
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - MD Anderson League City, League City, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Mary Washington Hospital, Fredericksburg, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - FHCC at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming